CLINICAL TRIAL: NCT06242717
Title: Postpartum Screening for Anxiety and Comorbid Conditions: A Prospective British Columbia Cohort Study
Brief Title: Postpartum Screening for Anxiety and Comorbid Conditions
Acronym: PPA
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Ministry of Health, British Columbia (Other Government); Providence Healthcare (Other); St. Paul's Hospital, Canada (Other); University of Victoria (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Marianne Vidler, Principle Investigator, University of British Columbia
Other Study IDs: H22-03298
Record Dates: First submitted 2023-11-08; First posted 2024-02-05 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Postpartum Anxiety; Postpartum Depression; Postpartum Disorder; Postoperative Pain; Sleep Wake Disorders; Quality of Life; Anger
MeSH Terms: conditions — Depression, Postpartum; Puerperal Disorders; Pain, Postoperative; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this project is to facilitate the design of individualized postpartum anxiety (PPA) screening strategies in British Columbia (BC), Canada. A cohort of postpartum people (n=550) will be invited to complete the following seven questionnaires at 4-8 weeks after delivery:

1. State-Trait Anxiety Inventory
2. Edinburgh Postnatal Depression Scale
3. Multidimensional Scale of Perceived Social Support
4. PROMIS (Patient-Reported Outcomes Measurement Information System) Emotional Distress-Anger, Short Form 5-a
5. Short Form Brief Pain Inventory
6. WHOQOL-BREF for assessing quality of life
7. PROMIS Sleep Disturbance Short Form 8-b and PROMIS Sleep-Related Impairment Short Form 8-a

The investigators will evaluate the feasibility of screening for postpartum anxiety and comorbid conditions through a web-based platform in a diverse BC population. They will assess the usability of the platform and questionnaires through 12-15 follow-up interviews with study participants and responses to the System Usability Scale. Their analysis will also identify patient characteristics and comorbidities (e.g., anger, pain, sleep disturbance) associated with a positive screen for postpartum anxiety.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 19 years
* 4-8 weeks postpartum
* Proficiency to participate in English
* Delivered within the province of British Columbia, Canada

Exclusion Criteria:

None.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cohort of postpartum people at 4-8 weeks after delivery.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who completed surveys | 4-8 weeks postpartum
  The overall completion rate will be estimated as those completing (defined as >70% completion rate) the entire screening divided by those recruited and will be provided with a corresponding 95% confidence interval.
Proportion of participants who consider usability of online surveys as being excellent (>85) with a System Usability Scale (SUS) | 4-8 weeks postpartum
  Feasibility will be determined by study completion rates and usability will be determined by SUS / b) SUS items have a range of 0-4. SUS scores range from 0 to 100 providing an estimate of overall usability of the intervention. Scores above 70 are considered to be acceptable or good while scores of 85 or above indicate a high level of usability or excellent score. Scores of 50 or below indicate poor or unacceptable usability. SUS scores and time to completion will be summarized based on above thresholds.

SECONDARY OUTCOMES:
Number of participants with postpartum-related anxiety as assessed by the State-Trait Anxiety Inventory (STAI-S) and related predictors. | 4-8 weeks postpartum
  A positive screen for anxiety will be determined using the validated questionnaire STAI (State-Trait Anxiety Inventory): 20-37 = No or Low Anxiety, 38-44 = "Moderate Anxiety", and 45-80 = "High Anxiety". / b) Possible predictors of a positive screen for anxiety will be initially assessed via summary statistics (e.g., mean differences or odds ratios) estimated via univariate regression models. / c) The investigators will assess the following predictors:
  Psychological risk factors: 1) "Past history of mood and/or anxiety disorders", 2) "Childhood abuse", 3) "Maternal sleep" / Biological risk factors: 1) "Proinflammatory T-helper cells and interleukins" / Obstetric and pregnancy-related factors: 1) "Difficult delivery", 2) "Negative obstetric outcomes", 3) "Current hyperemesis gravidarum", 4) "Breastfeeding" / Socio-demographic risk factors: 1) "Age", 2) "Marital status", 3) "Education level", 4) "Employment".
Number of participants with high postpartum-related anxiety and/or high risk for depression as assessed by validated questionnaires. | 4-8 weeks postpartum
  Common comorbidities that coincide with a positive screen for postpartum anxiety will be identified, as assessed by the STAI-validated questionnaire (as described in previous outcome measure) based on the responses to Edinburgh Postnatal Depression Scale (Range: 0-30, higher score: higher possibility of depression).
Number of participants with high postpartum-related anxiety and/or low social support as assessed by validated questionnaires. | 4-8 weeks postpartum
  Common comorbidities that coincide with a positive screen for postpartum anxiety will be identified, as assessed by the STAI-validated questionnaire (as described in previous outcome measure) based on the responses to Multidimensional Scale of Perceived Social Support Scale (Range: 12-84, lower score: lower social support).
Number of participants with high postpartum-related anxiety and/or high anger levels as assessed by validated questionnaires. | 4-8 weeks postpartum
  Common comorbidities that coincide with a positive screen for postpartum anxiety will be identified, as assessed by the STAI-validated questionnaire (as described in previous outcome measure) based on the responses to PROMIS Emotional Distress-Anger Short Form (5a, range: 5-25, higher score: more anger distress).
Number of participants with high postpartum-related anxiety and/or high levels of pain as assessed by validated questionnaires. | 4-8 weeks postpartum
  Common comorbidities that coincide with a positive screen for postpartum anxiety will be identified, as assessed by the STAI-validated questionnaire (as described in previous outcome measures) based on the responses to the Short Form Brief Pain Inventory Scale (Range: 0-120, higher score: higher pain severity).
Number of participants with high postpartum-related anxiety and/or low quality of life as assessed by validated questionnaires. | 4-8 weeks postpartum
  Common comorbidities that coincide with a positive screen for postpartum anxiety will be identified, as assessed by the STAI-validated questionnaire (as described in previous outcome measure) based on the responses to World Health Organization Quality of Life Scale (Range: 31-155, lower score: lower quality of life).
Number of participants with high postpartum-related anxiety and/or poor sleep quality as assessed by validated questionnaires. | 4-8 weeks postpartum
  Common comorbidities that coincide with a positive screen for postpartum anxiety will be identified, as assessed by the STAI-validated questionnaire (as described in previous outcome measure) based on the responses to PROMIS Sleep Disturbance (SF 8b) and Impairment (SF 8a) Scales (range: 16-80, higher score: more disturbed sleep).
Number of participants with two or more comorbid comorbidities as described on outcome measures 4 to 9. | 4-8 weeks postpartum
  Common comorbidities that coincide with a positive screen for postpartum anxiety will be identified, as assessed by the STAI-validated questionnaire (as described in previous outcome measure) based on the responses to validated questionnaires (as described in previous outcome measures). This will be done by estimating possible clusters of patients with commonalities. Cluster analysis based on hierarchical clustering will be conducted and assessed for internal validity via bootstrapping.

CONTACTS AND LOCATIONS:
Locations (1):
- BC Women's Hospital & Health Centre, Vancouver, British Columbia, Canada